CLINICAL TRIAL: NCT04385173
Title: A Pilot Study of Chimeric Antigen Receptor (CAR) T Cells Targeting B7-H3 Antigen in Treating Patients With Recurrent and Refractory Glioblastoma
Brief Title: Pilot Study of B7-H3 CAR-T in Treating Patients With Recurrent and Refractory Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: BoYuan RunSheng Pharma (Hangzhou) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU-BP102
Record Dates: First submitted 2020-02-04; First posted 2020-05-12 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Recurrent Glioblastoma; Refractory Glioblastoma
Keywords: Chimeric Antigen Receptor (CAR)-T; Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B7-H3 CAR-T (Experimental): Patients will received regular cycles of Temozolomide treatment with 5 days of treatment and 23 days of interval. 3 infusions of B7-H3 CAR-T with 1-2 weeks of interval will be used in between cycles of Temozolomide treatment. Temozolomide treatment during B7-H3 CAR-T infusions will be stopped and resumed after CAR-T infusion.
  Interventions: Drug: B7-H3 CAR-T; Drug: Temozolomide

INTERVENTIONS:
Drug: B7-H3 CAR-T — The B7-H3 CAR-T will be administrated via intratumoral or Intracerebroventricular injection through an Ommaya catheter in between Temozolomide cycles. Temozolomide will be stopped during the infusion of B7-H3 CAR-T
  Other Names: BP102
Drug: Temozolomide — Temozolomide will be given to patients orally every 5 days with 23 days interval. The initial dose is 150 mg/m2 on the first day and 200 mg/m2 for the rest if no toxicity is seen. If 200 mg/m2 is toxic, the drug will return to 150 mg/m2 or will be stopped.
  Other Names: TMZ

SUMMARY:
This is a pilot phase I study to evaluate the safety and efficacy on B7-H3 CAR-T in between Temozolomide cycles in treating patients with glioblastoma that has come back or does not respond to the standard treatment. The antigen B7-H3 is highly expressed in glioblastoma of a subset of patients. B7-H3 CAR-T, made from isolated patient peripheral blood mononuclear cells, can specifically attack patient glioblastoma cells that expressing B7-H3.

DETAILED DESCRIPTION:
Background

* B7-H3 is expressed in 70% of patients with glioblastoma
* B7-H3 is not expressed in normal tissues especially not in central nervous system. Therefore, it is an attractive GBM target for CAR-T therapy
* The investigators constructed a retroviral vector encoding a chimeric antigen receptor (CAR) targeting B7-H3, which can mediate CAR transfer into patient T cells with high efficiency.

Objectives

* To evaluate the safety and tolerability intratumoral/intracerebroventricular injection of B7-H3 CAR-T when used in between Temozolomide cycles
* To compare the overall survival (OS) and progression-free survival (PFS) of R/R GBM patients treated with B7-H3 CAR-T in between Temozolomide cycles to the historical Temozolomide data
* To access the pharmacokinetics and pharmacodynamics of B7-H3 CAR-T in between Temozolomide cycles

Design

Patients autologous T cells are activated and transduced with retrovirus containing B7-H3 CAR. CAR-T cells are expanded ex vivo and infused back to patients via intratumoral or intracerebroventricular injection through an Ommaya catheter. 3 injections of CAR-T are planned at two different doses with 1-2 weeks intervals. The CAR-T injections occur in between Temozolomide (TMZ) cycles. Temozolomide treatment in the cycle of CAR-T injections will be stopped and resumed next cycle. Patients may receive additional CAR-T cycles at the discretion of the principal investigator and oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.
* Histologically confirmed diagnosis of World Health Organization (WHO) classification grade IV glioblastoma (GBM).
* Clinical Pathology confirms B7-H3 positive tumor expression by immunohistochemistry (IHC) at the initial tumor presentation or recurrent disease (H-score >= 50).
* Relapsed/refractory disease confirmed by radiographic evidence after standard therapy.
* Suitable for the surgery of the placement of the Ommaya catheter.
* Eastern Cooperative Oncology Group (ECOG) =0 or 1 (need to be confirmed before intratumoral or intracerebroventricular injection)
* >= 8 weeks after completion of front-line radiation therapy
* >= 6 weeks after completion of nitrourea chemotherapy
* >= 14 days after completion of Temozolomide or other chemotherapy
* 2 weeks of wash-out time after completion of targeted therapy with related adverse events (AE) on baseline (4 weeks for Bevacizumab).
* Patients with other chronic AEs are in the investigator's judgement
* Blood cell count： White blood count (WBC) >= 2000/μL；Neutrophil count >= 1500/μL；Platelets >= 100 x 103/μL；Hemoglobin >= 9.0 g/dL
* Serum Creatinine <= 1.5×ULN or Creatinine Clearance Rate (Cockcroft and Gault) > 30 mL/min/1.73 m2
* Alanine Transaminase (ALT) <= 5×ULN and total bilirubin < 2.0mg/dL
* Lung function: Oxygen (O2) saturation >= 92% on room air and < CTCAE grade 1 dyspnea
* Heart function: Left ventricular ejection fraction (LVEF) >= 40% by multigated acquisition (MUGA) scan or echocardiogram
* Normal coagulation function: prothrombin time (PT)，activated partial thromboplastin time (APTT) and international normalized ratio (INR)
* Good blood vessel condition for leukapheresis
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity within one year after B7-H3 CAR-T infusion

Exclusion Criteria:

* Other active malignancy in the past 2 years except non-melanoma skin cancer, completely surgical removed low grade tumor, posttherapeutic limited-stage prostate cancer, biopsy confirmed in situ cervical carcinoma, PAP test confirmed squamous intraepithelial lesions
* Participant is undergoing or planning to take other anti-tumor therapies
* Participant is systematic steroid-dependent, or is expecting to be treated with systematic steroid
* Active immunodeficiency virus (HIV) or hepatitis B or hepatitis C virus infection
* Active infection from fungi, bacteria and/or viruses
* Known history of the following cardiac diseases in the past 6 months:
* New York Heart Association (NYHA) defined grade III or IV heart failure, cardiac angioplasty, myocardial infarction, unstable angina and other clinically significant heart diseases
* Known history and/or clinically evident central nerve system diseases: seizure, epileptic seizure, aphasia, paralysis, stroke, severe brain damage, dementia, Parkinson's Disease, cerebellar diseases, organic brain syndrome and psychiatric disorders
* Autoimmune diseases
* Pregnant or breastfeeding females
* Therapeutic doses of corticosteroid within 7 days before leukapheresis or 72 hours before B7-H3 CAR-T infusion
* Cytotoxic chemotherapy without lymphocytotoxicity within 1 week before leukapheresis except that the treatment has been stopped for more than 3 half-lives of the drug
* Lymphocytotoxic chemotherapy (cyclophosphamide, Ifosfamide and bendamustine) within 2 weeks before leukapheresis
* Other clinical trials drugs within 4 weeks before leukapheresis except that the drug has no effect or the disease has progressed, and the treatment has been stopped for more than 3 half-lives of the drug
* Radiotherapy within 6 weeks before leukapheresis
* Prior trials of CAR-T or other cell therapy
* Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of adverse events | 12 weeks
  Number of Participants With Treatment-Related Adverse Events and Types of adverse events as Assessed by CTCAE v4.0
Maximum tolerated dose (MTD) | 12 weeks
  The highest dose of B7-H3 CAR-T that does not cause targeted dose limiting toxicity
Overall survival (OS) | 2 years, up to 15 years if necessary
  Kaplan Meier methods will be used to estimate median OS
Progression-free survival (PFS) | 2 years, up to 15 years if necessary
  Kaplan Meier methods will be used to estimate median PFS. Progression is defined by Response Assessment in Neuro-Oncology (RANO) criteria

SECONDARY OUTCOMES:
The pharmacokinetics (PK) of B7-H3 CAR-T | 12 weeks
  Peak Concentration (Cmax) of B7-H3 CAR-T in peripheral blood (PB) and cerebral spinal fluid (CSF)
The pharmacokinetics (PK) of B7-H3 CAR-T | 12 weeks
  Area under the concentration versus time curve (AUC) of B7-H3 CAR-T in peripheral blood (PB) and cerebral spinal fluid (CSF)
Disease response (ORR, CR, PR, DOR) | 2 years, up to 15 years if necessary
  Objective Response Rate (ORR) will be assessed by comparison with baseline magnetic resonance imaging by RANO. Complete Response (CR) is disappearance of all measurable and non-measurable disease for at least 4 weeks. Partial Response (PR) is >/= 50% decrease in lesions for at least 4 weeks. Duration of Response (DOR) is the time between the initial response to the treatment and subsequent disease progression.

OTHER OUTCOMES:
Cytokine levels in PB and CSF | 12 weeks
  The concentration of cytokines (IL-1, IL-2, IL-6, IL-10, TNF-α, IFN-γ) in PB and CSF
T cell phenotype | 12 weeks
  The chimeric antigen receptor positive (CAR+) T cell and memory/effector T cell percentages and cell counts detected in peripheral blood (PB), and cerebral spinal fluid (CSF). Statistical and graphical methods will be used to describe persistence and expansion

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided